CLINICAL TRIAL: NCT00625794
Title: A Randomized Trial of the Nicotine Nasal Spray in Adolescent Smokers
Brief Title: Nicotine Replacement and Counseling In Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Mark Rubinstein, MD, UCSF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23RR018471 (NIH); 1K23RR018471 (NIH)
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2007-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 8 weeks or counseling plus 6 weeks of nicotine nasal spray
  Interventions: Drug: Nicotine nasal spray
- 2 (Active Comparator): 8 weeks or counseling only.
  Interventions: Behavioral: Smoking cessation counseling

INTERVENTIONS:
Drug: Nicotine nasal spray — 8 weeks or counseling plus 6 weeks of nicotine nasal spray (2 sprays each nostril as needed).
  Arms: 1
Behavioral: Smoking cessation counseling — 8 weeks or counseling
  Arms: 2

SUMMARY:
The objective of this pilot study is to determine the feasibility and utility of using the nicotine nasal spray (NNS) in adolescent smokers who want to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Be between 15 and 18 years-old
* Smoke 5 or more cigarettes per day (cpd) for at least 6 months and want to quit smoking.

Exclusion Criteria:

* Adolescents who were using or had used nicotine replacement in the prior week were excluded.
* Those who used bupropion (Zyban®) within the past 30 days were also excluded.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Self-reported smoking abstinence verified by both expired-air carbon monoxide and salivary cotinine. | 12 weeks

SECONDARY OUTCOMES:
Acceptability of the Nicotine Nasal Spray by Adolescents. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rubinstein, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States